CLINICAL TRIAL: NCT05068544
Title: Adolescent Normative Sport Movement Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/06/2
Record Dates: First submitted 2021-09-23; First posted 2021-10-06 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Lower Extremity Problem; Musculoskeletal Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to collect baseline data from a normative population of adolescents who participate in organized "land-based" sports, that gender and age matches some of the population of patients expected to be treated at Mary Bridge Children's Therapy Services, MultiCare affiliated therapy centers, and Mary Bridge Specialty Clinics who will be seen in the Research and Movement Lab. This project will recruit 40 patients between the ages of 13-25 years old. Non-invasive measurements of movement patterns will be collected during common sport-related activities over a single data collection session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13-25 years.
* Participate in a "land-based" organized sport in the last 1 year with intent on continued participation in the next year.
* Perform sport-related activities such as running/sprinting, cutting maneuvers, and jumping.
* Tolerate adhesive markers placed on skin and clothing.
* Willing and interested in participating.

Exclusion Criteria:

* Neuromuscular disorders such as cerebral palsy, muscular dystrophy, myotonic dystrophy, spinal muscular atrophy, peripheral neuropathy, or other generalized muscle and/or nerve issues.
* Currently undergoing treatment or receiving medication that affects movement.
* Requires ankle/knee bracing to safely perform running, sprinting, jumping activities.
* History of orthopedic surgery to lower limbs.
* In last 6 months: receiving/seeking medical treatment for injury.
* Difficulty performing sport-related activities.
* Pain that has inhibited participation in sports/daily activities in the last 3 months.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A group of 40 neurotypical and healthy adolescent subjects who participate in organized "land-based" sports will be recruited for this data collection. Adolescent subjects will be ages 13-25 with an equal number of male and female (gender assigned at birth).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Observation-based movement analyses | Baseline
  The purpose of the sports normative data collection is to develop a baseline database from a normative population of adolescents who participate in organized "land-based" sports. Observation-based analyses are performed with a trained practitioner identifying events (e.g. max knee flexion) and general joint position (e.g. knee valgus) through visual observation, or with the aid of video. This project will recruit 40 patients between the ages of 13-25 years old. Non-invasive measurements of movement patterns will be collected during common sport-related activities over a single data collection session.

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Bridge Children's Therapy Unit, Puyallup, Washington, United States

IPD SHARING:
Plan to Share IPD: No